CLINICAL TRIAL: NCT03543033
Title: Randomized Control Trial Comparing Pain and Functional Outcome Following Single Level Lumbar Nerve Decompression Surgery With or Without Preoperative Corticosteroid Epidural Injection
Brief Title: Preoperative Corticosteroid Epidural Injection and Lumbar Decompression Surgery Outcomes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was closed by the investigators due to lack of study population to enroll.
Sponsor: Lahey Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-008
Record Dates: First submitted 2018-04-11; First posted 2018-06-01 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Lumbar Radiculopathy
Keywords: lumbar radiculopathy; corticosteroid epidural injection
MeSH Terms: conditions — Radiculopathy | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial with randomization ratio 1:1
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Patients will receive a corticosteroid epidural injection within 2 weeks of their scheduled lumbar surgery
  Interventions: Drug: Corticosteroid injection
- Control (No Intervention): Patients will not receive a corticosteroid injection within 2 weeks of their scheduled lumbar surgery.

INTERVENTIONS:
Drug: Corticosteroid injection — These subjects will first receive a topical anesthesia to the skin and underlying tissue in a maximum amount of 5 ml of 1% Lidocaine. Following this application, an 18-20 gauge epidural needle will be used to inject a solution containing 80 mg Depo-Medrol in 1 ml of 1% PF Lidocaine and 5ml of sterile PF saline
  Arms: Treatment

SUMMARY:
This randomized control trial will compare opioid use, pain, and functional outcomes following decompression surgery for single-level lumbar radiculopathy in patients who undergo placement of corticosteroid epidural injection within 2 weeks prior to surgery compared to those who do not. The hypothesis of this study is that patients who receive the preoperative corticosteroid injection will have less reduced postoperative opioid use, as well as earlier mobilization, reduced length of stay, and faster return to work compared to control patients who do not receive the injection.

DETAILED DESCRIPTION:
This is a randomized control study that will be completed within the Department of Neurosurgery at Lahey Hospital & Medical Center. Patients will undergo their recommended surgery to treat single-level lumbar radiculopathy. Patients who are randomized to and consent to receiving a preoperative corticosteroid injection will report to clinic within 2 weeks prior to date of surgery to receive a corticosteroid injection. These subjects will first receive a topical anesthesia to the skin and underlying tissue in a maximum amount of 5 ml of 1% Lidocaine. Following this application, an 18-20 gauge epidural needle will be used to inject a solution containing 80 mg Depo-Medrol in 1 ml of 1% PF Lidocaine and 5ml of sterile PF saline. To assure the injection is epidural, we will be using loss of resistance technique under fluoroscopy and epidural placement will be confirmed with the live-image instillation in the AP and lateral positions of dye, with pattern confirming epidermal needle placement.

All patients will complete health outcome questionnaires (VAS, EQ-5D, ODI) at baseline (treatment cohort: prior to injection, control cohort: prior to spine surgery), 1 week post-op, 1 month post-op, and 3 months post-op. Patients will be instructed to bring all condition-related pain medication containers to each follow-up for research measuring purposes. Research personnel will record number of pills remaining in container, number of opioid prescription refills, and respective dates. Opioid usage for each subject will be tracked and converted to mg oral morphine equivalents using a standard table. Research personnel will capture additional clinic information such as length of stay, length of time before ambulation, and occurrence of any complications (i.e. DVT, infection). Opioid use, muscle relaxants, and other pain medication use will be followed for 3 months. At baseline and at each post-op follow up, patients will be asked to define their use of illicit drugs over the past 6 months (heroin, cocaine, marijuana, methamphetamine, other). Return to work date and work status will be captured out to 3 months. Patients will submit a health-cost diary at 1 week, 1 month, and 3 months, and this data will be combined with hospital-based cost information to generate a cost analysis. This diary will capture costs such as medication costs, copayments, travel, etc. Additionally, all patient surgery cancelations as well as reason for cancelation will be recorded. No additional medical testing will be required by the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 30-75 years of age
2. Patients diagnosed with diagnoses with single level unilateral lumbar radiculopathy
3. Patients diagnosed with spinal stenosis or disc herniation
4. Patients who have a history of > 6 weeks of at least 1 conservative treatment
5. ASA < III

Exclusion Criteria:

1. Patients who have undergone previous lumbar spinal surgery at index level
2. Patients diagnosed with spondylolisthesis at index level
3. Patients currently taking anti-coagulant therapy
4. Active treatment of major psychiatric condition such as major depression and/or anxiety disorder.
5. Patients currently seeking or receiving workers compensation
6. Patients who have undergone previous corticosteroid injection at index level
7. Morbid obesity defined as BMI > 40
8. Patients with history of chronic opioid use
9. Patients with a contrast dye allergy
10. Extruded disc fragment

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Opioid Use - conversion to oral morphine equivalents using standard table | Primary endpoint is 3 Months
  Following spine surgery, # of prescription opioid pills used will be recorded and converted to oral morphine equivalents using a standard table. Information collected will include # of pills taken, # of prescription refills, and respective dates.

SECONDARY OUTCOMES:
Disability - Oswestry Disability Index (ODI) | Baseline, 1 week post-op, 1 month post-op, and 3 months post-op
  Oswestry Disability Index (ODI) will be used to measure disability associated with their spinal condition. The ODI contains 10 questions; each with 6 choices and each answer choice ranges from 0 to 5 points. The minimum score is 0 and maximum score is 50; the higher the score, the greater the disability indicated. Each question is 5 points each and is summed then divided by total possible point. Scores from each cohort will be compared.
Pain - Visual Analog Scale (VAS) | Baseline, 1 week post-op, 1 month post-op, and 3 months post-op
  VAS will be used to measure pain and discomfort. The scale is a horizontal line numbered 0 through 10 with "0" indicating no pain, "5" indicating moderate pain, and 10 indicating worst pain. Patients will be instructed to mark an "X" on the number corresponding to their level of back pain over the past week. They will also be asked to indicate their leg pain on a similar, but separate scale. Scores from each cohort will be compared.
Quality of Life - EuroQol-5D | Baseline, 1 week post-op, 1 month post-op, and 3 months post-op
  EuroQol-5D (EQ-5D) will be used to measure quality of life. The EQ-5D includes 5 multiple-choice questions with 3 choices each; each choice corresponding to a value of 1,2,or 3. Each value is entered into an algorithm that computes a score. The score can range from "1" = high quality of life" and "0" = poor quality of life. Scores will be compared between both cohorts.

OTHER OUTCOMES:
Cost Analysis - Health Resource Diary | 1 week post-op, 1 month post-op, 3 months post-op
  A self-administered health resource diary will be completed by the patient. Information on co payments, travel costs, medical devices, and medical tests will be collected. Along with their estimated costs or receipts.

CONTACTS AND LOCATIONS:
Overall Officials: Erica J Bial, M.D., M.S., Principal Investigator — Lahey Clinic; Robert G Whitmore, M.D., Principal Investigator — Lahey Clinic
Locations (1):
- Lahey Hospital & Medical Center, Burlington, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No